CLINICAL TRIAL: NCT00390260
Title: Randomized, Double-Blind, Placebo-Controlled Trial of the Effect of Rofecoxib 50 mg and Hydrocodone 7.5 mg With Acetaminophen 750 mg in Patients With Postoperative Arthroscopic Pain
Brief Title: Effect of Rofecoxib and a Narcotic Analgesic to Treat Pain Following Arthroscopic Surgery (0966-179)(COMPLETED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0966-179; 2006_535
Record Dates: First submitted 2006-10-18; First posted 2006-10-19 (Estimated); Last update posted 2017-02-02 (Estimated); Status verified 2017-01

CONDITIONS: Pain, Postoperative Arthroscopy
MeSH Terms: conditions — Pain | interventions — rofecoxib; Duration of Therapy; Hydrocodone

INTERVENTIONS:
Drug: MK0966 / Duration of Treatment: 1 Days
Drug: Comparator: acetaminophen (+) hydrocodone bitartrate / Duration of Treatment: 1 Days
Drug: Comparator: placebo (unspecified) / Duration of Treatment: 1 Days

SUMMARY:
Study the effect of rofecoxib 50 mg compared to both placebo, and hydrocodone 7.5 mg with acetaminophen 750 mg, to treat moderate to severe pain following arthroscopic knee surgery.

ELIGIBILITY:
Inclusion Criteria:

* Elective outpatient arthroscopic knee surgery expected to last <= 90 minutes using general anesthesia
* Patients must experience moderate to severe pain following surgery
* Patient must be in general good health as judged by the primary investigator

Exclusion Criteria:

* Osteoarthritis; rheumatoid arthritis
* Allergy/sensitivity to aspirin, ibuprofen, indomethacin, other NSAIDs, COX-2 inhibitors (e.g., rofecoxib, celecoxib), hydrocodone, acetaminophen
* Asthma associated with nasal polyps
* Any arthroscopic knee surgery in the past 6 months

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 420
Dates: Start 2002-02; Primary Completion 2003-02 (Actual); Study Completion 2003-02 (Actual)

PRIMARY OUTCOMES:
Total Pain Relief over 6 hours following a single oral dose compared to placebo. | 6 hours

SECONDARY OUTCOMES:
Total Pain Relief over 6 hours following a single oral dose compared to hydrocodone + acetaminophen. | 6 hours

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Chelly JE, Nissen CW, Rodgers AJ, Smugar SS, Tershakovec AM. The efficacy of rofecoxib 50 mg and hydrocodone/acetaminophen 7.5/750 mg in patients with post-arthroscopic pain. Curr Med Res Opin. 2007 Jan;23(1):195-206. doi: 10.1185/030079907X162647. PMID 17207303
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/policies-perspectives.html